CLINICAL TRIAL: NCT01192308
Title: PharmacoKINEtics of TAMoxifen and Its Metabolites in Breast Cancer Patients: the Influence of a Dose Increase in Phenotypic Poor Metabolizers of CYP2D6 (KINETAM)
Acronym: KINETAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KINETAM
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Tamoxifen; Pharmacokinetics; Pharmacogenetics; CYP2D6
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 40mg QD dose intervention (Experimental): 40mg QD dose intervention during 4 weeks in patients with CYP2D6 variant allele or using CYP2D6 inhibitor.
  Interventions: Drug: Tamoxifen 40mg QD

INTERVENTIONS:
Drug: Tamoxifen 40mg QD — Tamoxifen 40mg QD during 4 weeks
  Other Names: Nolvadex

SUMMARY:
All women on tamoxifen receive the standard dose of 20mg QD, irrespective of the use of potential CYP2D6 inhibitors, and are not tested for CYP2D6 polymorphisms prior to start of tamoxifen treatment.However CYP2D6 polymorphisms and/or the use of CYP2D6 inhibitors as co-medication may influence the treatment outcome of tamoxifen.

The investigators propose a prospective study in women taking tamoxifen at a dose of 20mg QD. In each woman, information will be collected on endoxifen levels, CYP2D6 status, adherence and use of co-medication. In women who are phenotypically poor metabolizers of tamoxifen, a dose increase to 40mg QD will be applied and the effect of this intervention on tamoxifen pharmacokinetics will be evaluated after 4 weeks.

DETAILED DESCRIPTION:
Although already some information is available on the importance of CYP2D6 polymorphisms and/or the use of CYP2D6 inhibitors as co-medication that may influence the treatment outcome of tamoxifen, this information does currently not lead to a change in the management of this patient population. All women on tamoxifen receive the standard dose of 20mg QD, irrespective of the use of potential CYP2D6 inhibitors, and are not tested for CYP2D6 polymorphisms prior to start of tamoxifen treatment.

In an attempt to at least resolve some of these issues we propose a prospective study in women taking tamoxifen at a dose of 20mg QD who are being followed at several large oncology clinics in the south-eastern part of the Netherlands (Nijmegen (CWZ & Radboud), Den Bosch, Harderwijk and Arnhem). In each woman, information will be collected on endoxifen levels, CYP2D6 status, adherence and use of co-medication. In women who are phenotypically poor metabolizers of tamoxifen, a dose increase to 40mg QD will be applied and the effect of this intervention on tamoxifen pharmacokinetics will be evaluated after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years at screening.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is a female patient with (a history of) breast cancer and has been treated with tamoxifen 20mg QD for at least 4 weeks and is expected to be treated for at least another 4 weeks

Exclusion Criteria:

* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Tamoxifen and metabolites plasmaconcentration | week 0 and 4
  Trough samples

SECONDARY OUTCOMES:
Adverse events | week 0 and 4
  Collection of adverse events during entire trial.

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Result] Welzen ME, Dezentje VO, van Schaik RH, Colbers AP, Guchelaar HJ, van Erp NP, den Hartigh J, Burger DM, van Laarhoven HW. The Effect of Tamoxifen Dose Increment in Patients With Impaired CYP2D6 Activity. Ther Drug Monit. 2015 Aug;37(4):501-7. doi: 10.1097/FTD.0000000000000195. PMID 26192892